CLINICAL TRIAL: NCT02224885
Title: Needle-based Confocal Laser Endomicroscopy in Fluoroscopy-guided Procedures for Lung Applications (Biopsies and Ablation) and Liver Procedures in Interventional Radiology: a Feasibility Study
Brief Title: Needle-based Confocal Laser Endomicroscopy in Fluoroscopy-guided Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKT-IR-HEGP-2014
Record Dates: First submitted 2014-07-28; First posted 2014-08-25 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Lung Percutaneous Biopsy; Liver Percutaneous Biopsy
Keywords: Interventional radiology; Lung; Liver; Confocal endomicroscopy; Optical biopsy; Scanner; Fluoroscopy; CT; Computed Tomography; Radiofrequency Ablation; Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- addition of nCLE to help target biopsy (Other): The patient, scheduled for a liver or lung CT-guided percutaneous biopsy or ablation will undergo a probe-based confocal laser endomicroscopy procedure after the imaging procedure. The objectives of this study are to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure and determine whether it is technically feasible to obtain images from Cellvizio during an interventional radiology procedure.
  Interventions: Device: CT-guided percutaneous biopsy or ablation

INTERVENTIONS:
Device: CT-guided percutaneous biopsy or ablation — Standard interventional radiology procedure for a biopsy or ablation in the liver or in the lung

SUMMARY:
This study is a prospective study in order to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure in two main indications: lung and liver.

This innovative study will involve the use of probe-based confocal laser endomicroscopy. The proposed study is a feasibility study.

DETAILED DESCRIPTION:
Interventional radiology is a medical sub-specialty of radiology which utilizes minimally-invasive image-guided procedures to diagnose and treat diseases in nearly every organ. The concept behind interventional radiology is to diagnose and treat patients using less invasive techniques currently available in order to minimize risk to the patient and improve health outcomes.

For many years, surgery was the only treatment available for many conditions. Today, interventional radiology treatments are frst-line care for a wide variety of conditions. Patients should be offered the least invasive option frst. It is important to get a second opinion and know all of your treatment options before consenting to any procedure or surgery. Interventional radiologists are specialists in minimally invasive treatments, have a unique breadth of training and provide consults to every type of specialist.

Surgical removal of liver tumors offers the best chance for a cure. Unfortunately, liver tumors are often inoperable because the tumor may be too large, or has grown into major blood vessels or other vital structures. Sometimes, many small tumors are spread throughout the liver, making surgery too risky or impractical. Surgical removal is not possible for more than two-thirds of primary liver cancer patients and 90 percent of patients with secondary liver cancer.

The objectives of this study are to demonstrate the technical feasibility and safety of doing endomicroscopic imaging during interventional radiology procedure in two main indications: lung and liver.

The goal is to determine whether:

* Cellvizio insertion during the interventional procedure leads to change in known adverse events / serious adverse events rate during and one month after the procedure
* It is technically feasible to obtain images from Cellvizio during an interventional radiology procedure
* Cellvizio is a helpful assistance to increase the efficacy of biopsy which require to evaluate its accuracy eg. the predictive value of Cellvizio compared to pathology results.

Secondary goals are to assess:

* Benefit of spatial accuracy for the yield of the biopsy procedure and potential subsequent intervention, e.g. radiofrequency ablation.
* Regarding lung biopsies and lung ablation, potential increase of a database to refine image interpretation criteria with pathologists.
* In liver application, the goal is to build a database of images and define image interpretation criteria with pathologists to start image interpretation work.
* The predictive value of biopsies with Cellvizio assistance for lung or liver tumor biopsies.

For both applications, technical feedback from the physicians is expected on how they think the combined use of the devices could change the care path. E.g. a certain step in the workflow might become obsolete or the workflow could lead to fewer patient visits.

For the safety of this protocol, the use of endomicroscopy will not change in any way the patient management and standard procedure, including the diagnosis nor treatment decisions. All the adverse events / serious adverse events will be noted during the procedure and one week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have an interventional radiology procedure for needle-biopsy or radiofrequency ablation purposes in lung or in liver, 18 years or older.
* Only subjects who have provided written informed consent for the study can be included in the study.

Exclusion Criteria:

* Known allergy to fluorescein
* Previous life-threatening allergic reactions and known hypersensitivity to contrast media
* Pregnancy or breast-feeding
* History of cardio-pulmonary disease (including bronchial asthma)
* Restricted renal function
* Elderly with diabetes mellitus
* Patients under a beta-blockers treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Measure adverse events frequency in the use of mini probes on the tumor | Up to 1 week
  Assessment of the safety of inserting Cellvizio confocal miniprobe in the tumor (nor increase in bleeding or tumor cell dissemination) through the frequency, type and severity of adverse events

SECONDARY OUTCOMES:
Creation of image bank | Up to 6 months
  A frst creation of an atlas of endomicroscopic images obtained in interventional radiology in the liver - for the lung, the atlas established for peripheral lung nodules in bronchoscopy applications will serve as a reference and will be tested prospectively.
Yield of nCLE (needle-based confocal laser endomicroscopy)-targeted Fluoroscopy-guided biopsies | Up to 5 months
  Yield of nCLE (needle-based confocal laser endomicroscopy)-targeted Fluoroscopy-guided biopsies to assess improvements compared to standard of care from guidance function of the device combination.
Evaluation of potential benefits of the device combination | Up to 5 months
  Potential clinical, operational and financial benefits of the combination of Mauna Kea Technologies' endomicroscopic solution and Siemens' C-arm solution derived from the improved decision making for treatment of lung and liver lesions during the procedure (a clinical benefit could be fewer negative biopsies; an operational benefit could be one step fewer in the care path and a financial benefit could be a quicker diagnosis/treatment time, thus being able to release the patient earlier).
Assessment of accuracy and predictive value of interpretation criteria | Up to 5 months
  Evaluation of the predictive value of Cellvizio as an increasing tool of biopsy performance.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier PELLERIN, Principal Investigator — HEGP, Paris, France
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No